CLINICAL TRIAL: NCT04840121
Title: ADHESIORT - Personalizing Window of Implantation During Frozen Embryo Transfer
Brief Title: Personalizing Window of Implantation During Frozen Embryo Transfer
Acronym: AdhesioRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Ovo (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IIS - 1006
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Fertility

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in either the study group - AdhesioRT or in the control group - standard of care. All participants recruited, including the control group, will have the AdhesioRT biopsies performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group - AdhesioRT (Active Comparator): Prior to frozen embryo transfer, participants will proceed with the AdhesioRT test. Participants randomized in the study group will proceed with frozen embryo transfer cycle according window of implantation determined by AdhesioRT.
  Interventions: Diagnostic Test: AdhesioRT
- Control Group - Standard of Care (Active Comparator): Prior to frozen embryo transfer, participants will proceed with the AdhesioRT test. Participants randomized in the control group will proceed with the first frozen embryo transfer cycle as per standard of care. In the event of unsuccessful implantation (negative serum pregnancy test), participants will proceed with subsequent frozen embryo transfer cycle according to window of implantation determined by AdhesioRT.
  Interventions: Diagnostic Test: AdhesioRT

INTERVENTIONS:
Diagnostic Test: AdhesioRT — AdhesioRT, a novel diagnostic genetic assay, developed by ovo R&D scientists, helps to predict the endometrial receptivity and embryo implantation.

SUMMARY:
Embryo implantation is a crucial event in the establishment of a pregnancy. Although the clinical and culture conditions to obtain a "good quality" embryo are well advanced today, endometrial receptivity remains a major barrier in assisted reproductive techniques. Once a high-quality embryo is transferred, impaired uterine receptivity is believed to be one of the major reasons behind failure of the establishment of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 to 40 inclusive at the time of oocyte retrieval
* Prescription of a single frozen embryo transfer - substituted cycle protocol
* Participant has at least 2 vitrified good quality blastocysts

Exclusion Criteria:

* Women undergoing fertility preservation
* Stage IV severe endometriosis
* Severe malformation, adenomyosis or uterine anomaly including fibroids deforming the uterine cavity ≥ 5 cm
* Positive results of screening for either participant or partner for HIV antibodies, Hepatitis B (other than surface antibodies present after vaccination) or Hepatitis C

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Determination of appropriate window of implantation | 14 days after embryo transfer
  Comparison between standard frozen embryo transfer and personalized frozen embryo transfer using AdhesioRT to determine a successful window of implantation

SECONDARY OUTCOMES:
Rate of clinical pregnancy | 14 days after embryo transfer
  Blood test to determine if the embryo transfer was successful or not

CONTACTS AND LOCATIONS:
Overall Officials: Isaac-Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No